CLINICAL TRIAL: NCT06009380
Title: Effectiveness of Dual Task Training Versus Usual Care in Patients With Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: Effectiveness of Dual Task Training in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Fatih Ozden, Assistant Professor, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TDA Dual Task
Record Dates: First submitted 2023-08-15; First posted 2023-08-24 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Knee Arthroplasty; Rehabilitation
MeSH Terms: interventions — Physical Therapy Modalities; Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): In addition to the program given to the control group, the dual task program will be given to the study group progressively as previously stated (Silsupadol et al., 2006). These applications will be explained to the patients or their relatives face-to-face in the clinical environment after the initial evaluation and then sent and followed up by telerehabilitation method and patients will always have access to programs and education. In addition, both groups will be told that they can contact the researcher upon request.
  Interventions: Other: Physiotherapy and Rehabilitation
- Control Group (Active Comparator): The control group will receive the usual post-operative care of stretching lower extremity strengthening balance exercises activities of daily living recommendations.
  Interventions: Other: Physiotherapy and Rehabilitation

INTERVENTIONS:
Other: Physiotherapy and Rehabilitation — The control group will receive the usual post-operative care of stretching lower extremity strengthening balance exercises and activities of daily living recommendations. In addition to the program given to the control group, the dual task program will be given progressively to the study group.

SUMMARY:
This study was planned to investigate the effectiveness of usual care and dual task program in patients who underwent total knee arthroplasty surgery. It is aimed to evaluate pain intensity, disability level, mini mental status, coordination, reaction time and functional status of the patients. The study will be conducted with volunteer patients who are followed up by the Orthopedics and Traumatology outpatient clinic of Bursa Cekirge State Hospital and who have undergone total knee arthroplasty surgery. It is aimed to evaluate at least 26 patients for the study. The first evaluation will be performed 6 weeks post-operatively and the second evaluation will be performed 2 months after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Having undergone unilateral total knee arthroplasty surgery and being 6 weeks postoperative
* Participate in all necessary follow-up assessments
* 60 years of age or older
* Understand simple commands
* Signing the consent form

Exclusion Criteria:

* A previous history of total knee arthroplasty
* Presence of revision surgery
* Presence of severe osteoarthritis in the contralateral knee
* Severe acute metabolic neuromuscular and cardiovascular diseases
* Extreme obesity (bmi>35)
* Presence of malignancy
* Have any other orthopedic or neurological problem that may affect treatment and assessments
* Situations that prevent communication
* Lack of cooperation during the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Change from Baseline VAS at 8 weeks
  On a 10 cm straight line or numeric scale, the patient is asked to mark the pain they feel (0: no pain, 10: excruciating pain).
Knee Society Short Form (KSSF) | Change from Baseline KSSF at 8 weeks
  The scale is a 9-item measure developed to assess total knee arthroplasty patients' satisfaction, expectations, physical activities, and clinical and functional status in the preoperative and postoperative period, reported by both the physician and the patient.
Mini-Mental State Examination (MMSE) | Change from Baseline MMSE at 8 weeks
  The mini mental test is categorized under five main headings: orientation (10 points), recording memory (3 points), attention and calculation (5 points), recall (3 points) and language (9 points). The scale is scored out of a total of 30 points and has two different variants for educated and uneducated people. Traditionally, scores between 24 and 30 are considered normal. A score below 24 indicates cognitive impairment. 18-23 is considered as mild dementia, 12-17 as moderate dementia and below 12 as severe dementia.
Dual-Task Questionnaire (DTQ) | Change from Baseline DTQ at 8 weeks
  The questionnaire consists of 10 items and each question is rated out of 5 points (ranging from 0 "never" to 4 "very often" or N/A "not applicable"). The score obtained is the average score per question (i.e. total score/10 for the questionnaire).
Cognitive Timed Up and Go Test (CTUG) | Change from Baseline CTUG at 8 weeks
  Patients are first asked to stand up from a sitting position, walk 3 m at their normal speed, turn around, walk back to the chair and sit down. Walking aids are allowed. Patients are asked to perform this test while performing a cognitive dual task (subtract 2 continuously starting from 100).
Lower Extremity Motor Coordination Test (LEMCT) | Change from Baseline LEMCT at 8 weeks
  The test requires subjects sitting in a chair to alternately touch a proximal and distal target placed 30 cm apart on the floor with their feet within a 20-second period. A higher score indicates better motor coordination (13).
3 Meter Backward Walk Test (3MBWT) | Change from Baseline 3MBWT at 8 weeks
  A distance of 3 meters is measured and marked. Children are asked to walk backwards safely when the signal is given and stop when they reach the marked point. They are allowed to look behind them if necessary. Measurements are repeated 3 times and the average time is recorded.
10-Meter Walk Test (10MWT) | Change from Baseline 10MWT at 8 weeks
  A 10 meter long track is marked. Participants are instructed to "walk comfortably, at your usual pace" until they reach the end of the marked path. A member of the research team simultaneously measures the walking time with a stopwatch, starting the stopwatch as soon as the participant's lead foot crosses the first mark and stopping it when the participant's lead foot crosses the last mark. Distance and second data are used to determine walking speed.
Walking Impact Scale (Walk-12) | Change from Baseline Walk-12 at 8 weeks
  The test consists of 12 items asking about self-perceived walking limitations over the past 2 weeks in activities related to walking, running, climbing stairs, standing, walking distance and effort, need for support indoors and outdoors, elements of gait quality and concentration while walking. The scale has five response options: 1 = not at all, 2 = a little, 3 = moderately, 4 = somewhat and 5 = extremely. In clinical practice, the response options for each item are summed to obtain a total score ranging from 12 to 60 points.
Reaction Time Measurement (RTM) | Change from Baseline RTM at 8 weeks
  A platform with a circle on it is used to measure the stepping reaction. The participant standing outside the hoop is given a voice command and asked to step the relevant limb into the hoop. The time between immediately after the command and the first contact phase of stepping into the hoop is taken into account. The video images are evaluated with the Kinovea program using slow motion technology.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Özden, Study Director — Muğla Sıtkı Koçman University; Mustafa Yalçın, MSc, Principal Investigator — Bursa Çekirge State Hospital
Locations (1):
- Bursa Çekirge State Hospital, Bursa, Osmangazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No